CLINICAL TRIAL: NCT03255135
Title: Initial Experience in Brazilian Single Center With High Intensity Focalized Ultrasound (HIFU) Prostate Cancer Therapy: Morbidity, Oncological and Functional Outcomes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Transplante Doutor Euryclides de Jesus Zerbini (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU01
Record Dates: First submitted 2017-08-09; First posted 2017-08-21 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Transrectal High Intensity Focused Ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU (Experimental): Patients with untreated recent diagnosed localized prostate cancer candidates of focal therapy.
  Interventions: Device: HIFU

INTERVENTIONS:
Device: HIFU — High intensity focused ultrasound prostate cancer therapy guided by biopsy specimens and multiparametric prostate magnetic resonance using Focal One, Edap TMS, France device.

SUMMARY:
Prostate cancer (PCa) is the most prevalent non cutaneous cancer in occidental countries. In Brazil incidence was about sixty thousand new cases in 2016 and occupied second place as all cancer mortality, just behind lung cancer. Literature shows than younger patients tend to have more aggressive tumors rising cancer specific mortality scores. Main risk factors are age, life style (sedentary, high meat and fat intake) and family history (gene inheritance).

Besides vast advances in precocious tumors detection, challenges remain in the definition of the biological status of the tumor, which is highly variable and full of prognostic implications. PCa heterogeneity is demonstrated by the uncertain natural history, varying from indolent lesion to aggressive metastatic and fast progression cancer resistant to conventional therapies. In an actual treatment scenario, prognostic identification is the cornerstone of daily practice treatment considering the natural history variability cited before and the discrepancy of long term slow growth (studies estimate eight to sixteen years of tumor growth to achieve metastatic disease) to high grade aggressive cancer.

Considering all this background and taking in account the indolent evolution of low risk PCa new therapies emerge with promising outcomes. High-Intensity Focused Ultrasound (HIFU) have to be highlighted due to easy operation, good oncologic results and low complication profile. The method is based on real-time imaging guided high intensity ultrasound (US) causing overheat and cavitation in the focused tissue. Applied since 90's, mainly in German and French groups, initially programmed to treat hole gland preserving only urinary sphincter and bladder neck, showed recently some data on 1700 patients, 5 years biochemical recurrence free survival of 80% and best results including morbidity profile in low risk, low prostate volume and in the group with previous trans urethral prostate resection (TURP). This results are very similar to other radical treatment options with median follow up of 8 years, cancer specific survival 98% and metastasis free survival of 95% If local recurrence was identified another HIFU ablation or even radical treatment achieved good results in local control with acceptable morbidity profile.

Focal treatment is a new entity in PCa therapy. One randomized trial compared focal treatment to active surveillance in 513 mans with PCa diagnosis. With a 24 month follow-up progression-free ratios (28% x 58%) and positive control prostate biopsy ratios (14% x 49%) were fairly superior in treatment group. This exiting novel data turns urological oncology paths to the new era of minimally harmful therapy with targeted focused procedure. At our knowledge there is no high evidence clinical trial comparing HIFU to active surveillance.

The objective of this study is to evaluate prospectively the initial experience with 50 patients submitted to HIFU therapy for low risk prostate cancer in Brazilian single center considering the following aspects:

One year of treatment prostate biopsy positiveness; Biochemical recurrence free survival using Phoenix and Stuttgart criteria in one year; Sexual function using IIEF-5 questionnaire and the usage of 5-phosphodiesterase inhibitors (5-PDI); Urinary symptoms using EPIC and IPSS questionnaires and free urinary flow; Quality of life based on SF-36 questionnaire evaluation; Post procedure morbidity using Clavien-Dindo classification.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most prevalent non cutaneous cancer in occidental countries. In Brazil incidence was about sixty thousand new cases in 2016 and occupied second place as all cancer mortality, just behind lung cancer. Literature shows than younger patients tend to have more aggressive tumors rising cancer specific mortality scores. Main risk factors are age, life style (sedentary, high meat and fat intake) and family history (gene inheritance).

Screening programs suggested by urological and oncologic societies, mainly based on Prostate Specific Antigen (PSA), changed natural history of this disease, overturning past late diagnosis with advanced disease to early discover in present days, with localized highly curable cancer by local therapy (surgery or radiation therapy) turning focus on morbidity status based on the high long term cancer specific survival.

Besides vast advances in precocious tumors detection, challenges remain in the definition of the biological status of the tumor, which is highly variable and full of prognostic implications. PCa heterogeneity is demonstrated by the uncertain natural history, varying from indolent lesion to aggressive metastatic and fast progression cancer resistant to conventional therapies. In an actual treatment scenario, prognostic identification is the cornerstone of daily practice treatment considering the natural history variability cited before and the discrepancy of long term slow growth (studies estimate eight to sixteen years of tumor growth to achieve metastatic disease) to high grade aggressive cancer.

Aiming to reduce PCa cancer specific mortality, PSA tests associated with digital rectal examination are the actual standard of care in PCa screening. A randomized clinical trial demonstrated reduction in the risk of PCa death up to 25% in patients maintaining regular screening. Risk stratification after tumor diagnosis includes nomograms, most used is D'Amico score stratifying low, intermediate and high risk cancer based on PSA value, digital rectal examination, tumor histology and volume. Considering the risk, treatment may be localized, systemic or active surveillance.

Three randomized trials compared active surveillance with local treatment, one showing benefit in cancer specific survival with 40% reduction and other two demonstrating comparable outcomes. Considering this studies results, one important detail was related to metastasis, pointing that metastasis free survival was better for the treatment group compared to surveillance. Based on this studies active surveillance was introduced in guidelines and clinical practice with the benefits of minimizing morbidity and disadvantage of slightly higher risk of metastasis and local complications.

Radical prostatectomy (RP) have high cure rates, overall survival of 99% and cancer specific survival superior to 80%, however, deem to have quality of life changing implications that are at least relevant in this highly curable scenario. Urinary incontinence ranging from 1-15% and erectile dysfunction compromising about 40% of the patients (highly variable considering previous status, age, comorbidities, local and technical aspects) Radiation therapy is implied with slightly higher local recurrence when compared to RP, lower incontinence risk but can damage surrounding structures like bladder and rectum causing bothersome and difficult to manage bleeding (radiation cystitis and radiation proctitis can occur in 10 to 20% of patients). In intermediate or high risk groups radiation therapy alone has inferior oncologic results and is associated with periodic androgen deprivation therapy (ADT), aggregating other undesired effects (erectile dysfunction, osteopenia, muscular loss and cardiovascular disease).

Considering all this background and taking in account the indolent evolution of low risk PCa new therapies emerge with promising outcomes. High-Intensity Focused Ultrasound (HIFU) have to be highlighted due to easy operation, good oncologic results and low complication profile. The method is based on real-time imaging guided high intensity ultrasound (US) causing overheat and cavitation in the focused tissue. Applied since 90's, mainly in German and French groups, initially programmed to treat hole gland preserving only urinary sphincter and bladder neck, showed recently some data on 1700 patients, 5 years biochemical recurrence free survival of 80% and best results including morbidity profile in low risk, low prostate volume and in the group with previous trans urethral prostate resection (TURP). This results are very similar to other radical treatment options with median followup of 8 years, cancer specific survival 98% and metastasis free survival of 95% If local recurrence was identified another HIFU ablation or even radical treatment achieved good results in local control with acceptable morbidity profile.

HIFU morbidity profile seems acceptable when compared to the other treatments available. Urinary incontinence was mostly minor in 1-3%, sexual dysfunction compromised about 50% of the cases, urethral or bladder neck stricture in 5%. To reach this results, cancer centers associated TURP before HIFU ablation and optimized patient selection to reach the best of the method.

In 2014 the US Food and Drug Administration (FDA) approved HIFU use in prostate tissue ablation, hissing interest in this technology. Up to now 50 thousand patients undergone prostate ablation with HIFU (half of them to treat PCa). Recently some centers concentrated their efforts to establish focal treatment for PCa in detriment to hole gland. Focal treatment seems a good alternative to active surveillance and for a specific group of patients who are not candidates do radical therapy due to performance status, comorbidities or personal preferences.

In recent reports about prostate cancer biology, the index lesion seems to be the main therapy target due to aggressive comportment and higher dissemination potential, different from the secondary lesions that have indolent growth. Considering this paradigm, treat the index lesion seems to be a logical way to have good oncologic control with the best treatment related morbidity status, and is properly possible due to advances in radiologic imaging diagnosis using multi-parametric prostate magnetic resonance.

Focal treatment is a new entity in PCa therapy. One randomized trial compared focal treatment to active surveillance in 513 mans with PCa diagnosis. With a 24 month follow-up progression-free ratios (28% x 58%) and positive control prostate biopsy ratios (14% x 49%) were fairly superior in treatment group. This exiting novel data turns urological oncology paths to the new era of minimally harmful therapy with targeted focused procedure. At our knowledge there is no high evidence clinical trial comparing HIFU to active surveillance.

OBJECTIVE To evaluate prospectively the initial experience with 50 patients submitted to HIFU therapy for low risk prostate cancer in Brazilian single center.

The research team will evaluate:

1. One year of treatment prostate biopsy positiveness;
2. Biochemical recurrence free survival using Phoenix and Stuttgart criteria in one year;
3. Sexual function using IIEF-5 questionnaire and the usage of 5-phosphodiesterases inhibitors (5-PDI);
4. Urinary symptoms using EPIC and IPSS questionnaires and free urinary flow;
5. Quality of life based on SF-36 questionnaire evaluation;
6. Post procedure morbidity using Clavien-Dindo classification.

METHODS Patients selection will involve males with recent diagnosis of usual acinar prostate adenocarcinoma with Gleason score ranging from 6 to 7 (ISUP 1, 2 or 3). Maximum PSA level cutoff will be 15 with no minimum level. Digital rectal examination demonstrating organ confined cancer (clinical stage ≤T2c). There will be no limit on patients age and study candidates may not have been submitted to any Cap treatment. Other exclusion criteria will be rectal functional or anatomical abnormalities.

After patient entrance by study therm signature, there will be the first medical evaluation with medical history, full physical examination including digital rectal examination and pre-treatment questionnaires application (IIEF-5, EPIC, IPSS, SF-36). General blood samples, free urinary flow and any other examination that will be considered necessary by the assistant urologist will be collected in the first day of evaluation. Clinical and demographic data will be collected: age, symptoms, post-treatment complications, comorbidities, medications in use, previous surgery, alcohol, tobacco and other drugs usage, weight, height, blood count, urea, creatinine, C reactive protein, PSA (total and free portion), urine analysis and culture, urinary tract ultrasound, prostate ultrasound (US) with estimated prostate weight, multi-parametric prostate MRI (when feasible) considering PIRADs category, extra-prostatic extension, seminal vesicle compromising and lymph node status, presence of median lobe of prostate, bone scan (if indicated), number of biopsies fragments, positiveness of fragments, Gleason grade, tumor localization, percentage of tumor compromising in the fragment, need of previous TURP, bladder catheter usage, free urinary flow after TURP, pathology evaluation of TURP product, HIFU treatment time, HIFU treatment protocol (hole gland, half-gland or focal treatment), in hospital stay, time of urethral catheter usage, analgesics usage, opioids usage and post treatment questionnaires (IIEF-5, EPIC, IPSS e SF-36).

TREATMENT DESCRIPTION Procedures will take place in single reference urological hospital in Sao Paulo Brazil, with FocalOneR, Edap TMS, France as the device. Treatment will be planned in accordance with biopsy laterality in half-gland protocols for unilateral disease and whole gland ablation for bilateral cases. Neurovascular bundle preservation will occur on the contralateral side of the disease. Urinary sphincter margin will be planned with 3 millimeter distance to ensure sphincter preservation.

Every patient with prostate gland volume higher than 40 cc in pre-treatment US or MRI must have an TURP before ablation. In symptomatic patients with prostate volume lower than 40 cc assistant urologist clinical judgement will decide between doing or not pre-ablation TURP.

Rectal cleansing with enema is done up to 3 hours before procedure. Prophylactic antibiotic of choice is second generation cephalosporin (Cefuroxime 1.5 g intravenous), used 30 minutes before procedure.

Prostate cancer ablation will follow previous established treatment protocol from FocalOne: general anesthesia, Foley bladder catheter 16 or 18 Fr is inserted just before treatment and maintained up to 72 hours (Hole gland).

Post ablation medications includes antibiotics and analgesics if necessary. Patient discharge can take place at same ablation day if procedure finish up to 1 PM, otherwise patient discharge normally happen in first post-procedure day. Patients discharged with bladder catheter are orientated to return in ambulatory to take it off up to the third day after ablation.

FOLLOW UP First follow up medical visit occurs with 15 days after HIFU. Medical interview will focus on complications and adverse events. Follow up will continue with medical visits in 3, 6 and 12 months after procedure.

Evaluations in the follow up visits consist in clinical and physical examinations, digital prostate examination, obtainment of blood samples (PSA). When reaching 12 months after treatment patients will take another saturation prostate biopsy (20 fragments) for treatment control. Questionnaires IIEF-5, EPIC, IPSS, SF-36 and free urinary flow will be done at all medical visits (3, 6 e 12 months).

1. Post HIFU medical visits will occur at 3, 6 e 12 months;
2. First post ablation visit will occur at the 15th day;
3. Medical interview, physical examination with digital rectal prostate examination and blood sample obtain to PSA analysis will be collected in each of the medical visit except the PSA collection at 15th day one.
4. 12 months after treatment patients will take another saturation prostate biopsy (20 fragments) for treatment control;
5. Questionnaires IIEF-5, EPIC, IPSS, SF-36 and free urinary flow will be done at all medical visits (3, 6 e 12 months);

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with recent diagnosis of usual adenocarcinoma of prostate untreated and with indication of specific treatment by the assisting urologist;
* 2. And low or intermediate prostate cancer in clinical staging;
* 3. And concordance with the clinical trial by signing the terms.

Exclusion Criteria:

* 1. Other types of prostate cancer not usual adenocarcinoma;
* 2. Or any previous treatment to prostate cancer;
* 3. Or any patient who presents with proctologic abnormalities;

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer biochemical recurrence free survival after prostate cancer focal therapy | 12 months
  Biochemical recurrence free survival using Phoenix criteria in one year
Prostate cancer pathological persistence after prostate cancer focal therapy | 12 months
  One year post-HIFU treatment prostate biopsy positivity

SECONDARY OUTCOMES:
IIEF-5 - Sexual function after prostate cancer focal therapy | 12 months
  Sexual function using IIEF-5 questionnaire
5-PDI - Sexual function after prostate cancer focal therapy | 12 months
  Sexual function using evaluation of usage of 5-Phosphodiesterase inhibitors (5-PDI)
Free urinary flow - Urinary symptoms after prostate cancer focal therapy | 12 months
  Urinary symptoms using free urinary flow measure
EPIC - Urinary symptoms after prostate cancer focal therapy | 12 months
  Urinary symptoms using EPIC questionnaire
IPSS - Urinary symptoms after prostate cancer focal therapy | 12 months
  Urinary symptoms using IPSS questionnaire
Quality of life after prostate cancer focal therapy | 12 months
  Quality of life based on SF-36 questionnaire evaluation
Morbidity after prostate cancer focal therapy | 12 months
  Post procedure morbidity using Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Transplantes Euryclides de Jesus Zerbini, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Popiolek M, Rider JR, Andren O, Andersson SO, Holmberg L, Adami HO, Johansson JE. Natural history of early, localized prostate cancer: a final report from three decades of follow-up. Eur Urol. 2013 Mar;63(3):428-35. doi: 10.1016/j.eururo.2012.10.002. Epub 2012 Oct 13. PMID 23084329
- [Background] Gotoh M, Kondo A, Miyake K. Bladder compliance in myelodysplastic children: does antireflux surgery compromise it? Urol Int. 1991;47 Suppl 1:63-6. doi: 10.1159/000282253. PMID 1949380
- [Background] Jemal A, Ward EM, Johnson CJ, Cronin KA, Ma J, Ryerson B, Mariotto A, Lake AJ, Wilson R, Sherman RL, Anderson RN, Henley SJ, Kohler BA, Penberthy L, Feuer EJ, Weir HK. Annual Report to the Nation on the Status of Cancer, 1975-2014, Featuring Survival. J Natl Cancer Inst. 2017 Sep 1;109(9):djx030. doi: 10.1093/jnci/djx030. PMID 28376154
- [Background] Carter HB, Pearson JD. Prostate-specific antigen testing for early diagnosis of prostate cancer: formulation of guidelines. Urology. 1999 Nov;54(5):780-6. doi: 10.1016/s0090-4295(99)00271-x. No abstract available. PMID 10565733
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Zappa M, Nelen V, Kwiatkowski M, Lujan M, Maattanen L, Lilja H, Denis LJ, Recker F, Paez A, Bangma CH, Carlsson S, Puliti D, Villers A, Rebillard X, Hakama M, Stenman UH, Kujala P, Taari K, Aus G, Huber A, van der Kwast TH, van Schaik RH, de Koning HJ, Moss SM, Auvinen A; ERSPC Investigators. Screening and prostate cancer mortality: results of the European Randomised Study of Screening for Prostate Cancer (ERSPC) at 13 years of follow-up. Lancet. 2014 Dec 6;384(9959):2027-35. doi: 10.1016/S0140-6736(14)60525-0. Epub 2014 Aug 6. PMID 25108889
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Bill-Axelson A, Holmberg L, Garmo H, Rider JR, Taari K, Busch C, Nordling S, Haggman M, Andersson SO, Spangberg A, Andren O, Palmgren J, Steineck G, Adami HO, Johansson JE. Radical prostatectomy or watchful waiting in early prostate cancer. N Engl J Med. 2014 Mar 6;370(10):932-42. doi: 10.1056/NEJMoa1311593. PMID 24597866
- [Background] Wilt TJ, Brawer MK, Jones KM, Barry MJ, Aronson WJ, Fox S, Gingrich JR, Wei JT, Gilhooly P, Grob BM, Nsouli I, Iyer P, Cartagena R, Snider G, Roehrborn C, Sharifi R, Blank W, Pandya P, Andriole GL, Culkin D, Wheeler T; Prostate Cancer Intervention versus Observation Trial (PIVOT) Study Group. Radical prostatectomy versus observation for localized prostate cancer. N Engl J Med. 2012 Jul 19;367(3):203-13. doi: 10.1056/NEJMoa1113162. PMID 22808955
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Klotz L, Vesprini D, Sethukavalan P, Jethava V, Zhang L, Jain S, Yamamoto T, Mamedov A, Loblaw A. Long-term follow-up of a large active surveillance cohort of patients with prostate cancer. J Clin Oncol. 2015 Jan 20;33(3):272-7. doi: 10.1200/JCO.2014.55.1192. Epub 2014 Dec 15. PMID 25512465
- [Background] Bianco FJ Jr, Scardino PT, Eastham JA. Radical prostatectomy: long-term cancer control and recovery of sexual and urinary function ("trifecta"). Urology. 2005 Nov;66(5 Suppl):83-94. doi: 10.1016/j.urology.2005.06.116. PMID 16194712
- [Background] Wallis CJD, Saskin R, Choo R, Herschorn S, Kodama RT, Satkunasivam R, Shah PS, Danjoux C, Nam RK. Surgery Versus Radiotherapy for Clinically-localized Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2016 Jul;70(1):21-30. doi: 10.1016/j.eururo.2015.11.010. Epub 2015 Dec 15. PMID 26700655
- [Background] Gelet A, Chapelon JY, Bouvier R, Souchon R, Pangaud C, Abdelrahim AF, Cathignol D, Dubernard JM. Treatment of prostate cancer with transrectal focused ultrasound: early clinical experience. Eur Urol. 1996;29(2):174-83. PMID 8647143
- [Background] Thuroff S, Chaussy C. Evolution and outcomes of 3 MHz high intensity focused ultrasound therapy for localized prostate cancer during 15 years. J Urol. 2013 Aug;190(2):702-10. doi: 10.1016/j.juro.2013.02.010. Epub 2013 Feb 13. PMID 23415962
- [Background] Crouzet S, Chapelon JY, Rouviere O, Mege-Lechevallier F, Colombel M, Tonoli-Catez H, Martin X, Gelet A. Whole-gland ablation of localized prostate cancer with high-intensity focused ultrasound: oncologic outcomes and morbidity in 1002 patients. Eur Urol. 2014 May;65(5):907-14. doi: 10.1016/j.eururo.2013.04.039. Epub 2013 Apr 30. PMID 23669165
- [Background] van Velthoven R, Aoun F, Marcelis Q, Albisinni S, Zanaty M, Lemort M, Peltier A, Limani K. A prospective clinical trial of HIFU hemiablation for clinically localized prostate cancer. Prostate Cancer Prostatic Dis. 2016 Mar;19(1):79-83. doi: 10.1038/pcan.2015.55. Epub 2015 Nov 24. PMID 26597660
- [Background] Feijoo ER, Sivaraman A, Barret E, Sanchez-Salas R, Galiano M, Rozet F, Prapotnich D, Cathala N, Mombet A, Cathelineau X. Focal High-intensity Focused Ultrasound Targeted Hemiablation for Unilateral Prostate Cancer: A Prospective Evaluation of Oncologic and Functional Outcomes. Eur Urol. 2016 Feb;69(2):214-20. doi: 10.1016/j.eururo.2015.06.018. Epub 2015 Jul 9. PMID 26164416
- [Background] Ahmed HU. The index lesion and the origin of prostate cancer. N Engl J Med. 2009 Oct 22;361(17):1704-6. doi: 10.1056/NEJMcibr0905562. No abstract available. PMID 19846858
- [Background] Azzouzi AR, Vincendeau S, Barret E, Cicco A, Kleinclauss F, van der Poel HG, Stief CG, Rassweiler J, Salomon G, Solsona E, Alcaraz A, Tammela TT, Rosario DJ, Gomez-Veiga F, Ahlgren G, Benzaghou F, Gaillac B, Amzal B, Debruyne FM, Fromont G, Gratzke C, Emberton M; PCM301 Study Group. Padeliporfin vascular-targeted photodynamic therapy versus active surveillance in men with low-risk prostate cancer (CLIN1001 PCM301): an open-label, phase 3, randomised controlled trial. Lancet Oncol. 2017 Feb;18(2):181-191. doi: 10.1016/S1470-2045(16)30661-1. Epub 2016 Dec 20. PMID 28007457
- [Background] Rischmann P, Gelet A, Riche B, Villers A, Pasticier G, Bondil P, Jung JL, Bugel H, Petit J, Toledano H, Mallick S, Rouviere O, Rabilloud M, Tonoli-Catez H, Crouzet S. Focal High Intensity Focused Ultrasound of Unilateral Localized Prostate Cancer: A Prospective Multicentric Hemiablation Study of 111 Patients. Eur Urol. 2017 Feb;71(2):267-273. doi: 10.1016/j.eururo.2016.09.039. Epub 2016 Oct 6. PMID 27720531
- [Background] Ahmed HU, Hindley RG, Dickinson L, Freeman A, Kirkham AP, Sahu M, Scott R, Allen C, Van der Meulen J, Emberton M. Focal therapy for localised unifocal and multifocal prostate cancer: a prospective development study. Lancet Oncol. 2012 Jun;13(6):622-32. doi: 10.1016/S1470-2045(12)70121-3. Epub 2012 Apr 17. PMID 22512844
- [Background] Barret E, Ahallal Y, Sanchez-Salas R, Galiano M, Cosset JM, Validire P, Macek P, Durand M, Prapotnich D, Rozet F, Cathelineau X. Morbidity of focal therapy in the treatment of localized prostate cancer. Eur Urol. 2013 Apr;63(4):618-22. doi: 10.1016/j.eururo.2012.11.057. Epub 2012 Dec 13. PMID 23265382